CLINICAL TRIAL: NCT04950413
Title: Effect of Instrument-assisted Soft Tissue Mobilization and Phonophoresis on Trigger Points of Tension Headache
Brief Title: Instrument-assisted Soft Tissue Mobilization and Phonophoresis on Trigger Points of Tension Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nada Gamal Saad (Other)
Responsible Party: Sponsor-Investigator, Nada Gamal Saad, Sponsor Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nada_MSc
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Headache; Tension-Type Headache
MeSH Terms: conditions — Headache; Tension-Type Headache | interventions — Phonophoresis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional Treatment Arm (Active Comparator): conventional physical therapy program (infrared, stretching exercise, isometric strengthening exercise)
  Interventions: Other: Conventional physical therapy program
- IASTM treatment arm (Experimental): Instrument-assisted soft tissue mobilization (IASTM) is a therapeutic technique that is based on the soft tissue mobilization rationale introduced by James Cyriax.
  Interventions: Other: Conventional physical therapy program; Other: IASTM by M2t blade
- Phonophoresis treatment arm (Experimental): It will be consisted of 1 MHz pulsed mode with an intensity set at 1.5 W/cm2.
  Interventions: Other: Conventional physical therapy program; Device: Phonophoresis
- Combined IASTM and phonophoresis treatment arm (Experimental): Combined phonophoresis and M2t Blade
  Interventions: Other: Conventional physical therapy program; Other: IASTM by M2t blade; Device: Phonophoresis

INTERVENTIONS:
Other: Conventional physical therapy program — Infrared, Exercises, Stretching exercise of Suboccepital muscle
Other: IASTM by M2t blade — A lubricant (Vaseline) will be applied to the skin around the neck area prior to treatment and the M2t blade will be cleaned with an alcohol pad. First, the M2T blade will used to ﬁnd the exact areas of restriction in affected muscles. Then the M2T blade will use at an angle of 45 to apply slow strokes along the muscle. Changes in soft tissue consistency will detected by the clinician through vibrations of the instrument when it slides on areas of irregular fibrosis of the underneath connective tissue. Once an adhesion is discovered, strokes are repeated for 5 min.
  Arms: Combined IASTM and phonophoresis treatment arm; IASTM treatment arm
Device: Phonophoresis — It will be consisted of 1 MHz pulsed mode with an intensity set at 1.5 W/cm2 and. A 5 cm2 crystal head with an effective radiating area of 4.0 cm2 ±1.0 wills utilized for 5 Min for each trigger point of neck. lidocine gelwill applied instead of coupling US gel used for transmission.
  Arms: Combined IASTM and phonophoresis treatment arm; Phonophoresis treatment arm

SUMMARY:
General purpose:

It was investigate the effect of IASTM and phonophoresis on Tension Type headache.

Specific Purpose:

1. It was investigate the effect of IASTM on headache frequency, PPT, pain intensity, and functional disability on trigger points of tension type headache.
2. It was investigate the effect of Lidocaine phonophoresis on headache frequency, PPT, pain intensity and functional disability on trigger points of tension type headache.
3. It was investigate the effect of IASTM and Lidocaine phonophoresis on headache frequency, PPT, pain intensity, and functional disability on trigger points of tension type headache.

DETAILED DESCRIPTION:
Phonophoresis is the use of therapeutic ultrasound to increase percutaneous drug absorption Percutaneous administration offers many benefits such as steady plasma levels, lack of degradation by the gastrointestinal system, and lack of liver effects (first-pass drug metabolism) on drug molecules. Transdermal drug delivery offers a unique opportunity for non-invasive and controlled drug delivery, in contrast to needle-based and oral drug administration. Phonophoresis is a therapeutic method that may be helpful for the treatment of MTP.

There are potentially adverse treatment responses to ISTM that may occur. The patient may experience discomfort during the administration of the treatment, and petechiae (i.e., bruising) may become apparent during or after the treatment Although discomfort may be experienced, patients who have realized a decrease in symptoms have returned repeatedly for additional ISTM sessions other therapeutic modalities should be administered for pain management.

Clinical and scientiﬁc evidence supports that proper management of patients with headache should be multimodal including appropriate use of pharmacological and non-pharmacological.IASTM used to facilitate normal alignment of soft tissue and increase fibroblast recruitment and regeneration of damaged tissue. Phonophoresis is frequently used to treat pain associated with muscular disorders, enhancing skin absorption of the topical medication's molecules. Study report that lidocaine decreases sensory input from mrofascialTrps and release local Tenderness by lowering the degree of the reflex mechanism responsible for referred pain.

ELIGIBILITY:
Inclusion Criteria:

* Their age ranged from 30 to 40 years.
* BMI ranged from 18 to 25 kg /m2.
* TTH criteria according to the Headache Classification Committee of the International Headache Society has at least two of the following characteristics:
* Bilateral location.
* Pressing/tightening quality (non-pulsating).
* Mild or moderate intensity.
* Not aggravated by routine physical activity such as walking or climbing stairs.
* Patients have Trigger points in suboccipital muscle and trigger points 1 trapezius muscle.
* The presence of MTrPs will be determined using the diagnostic criteria described by Simons 1990, in which five major criteria and at least one of three minor criteria are needed for a clinical diagnosis of MPS.

Exclusion Criteria:

* Patients with a history of malignancy.
* Patients who had a history of cervical and cranial Surgery.
* Patients with major psychiatric disorders (major Depression).
* Patients with uncontrolled hypertension
* Patient with other causes of headache.
* Dysfunctions in the temporomandibular joint.
* Headaches associated with high fever, stiff neck, or rash, problems with vision, or profound dizziness.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Assessing the change in pain intensity | Baseline and 4 weeks post-intervention
  assessment via using visual analogue scale (VAS) most commonly consists of a 100mm horizontal line anchored with two opposite labels; patients mark a score on the scale using a vertical line. A VAS is easy to use and therefore applicable to a variety of practice and research settings. (0 means no pain & 10 means highest pain intensity).
Assessing the change in neck disability | Baseline and 4 weeks post-intervention
  assessment via using Neck disability index: The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means: no activity limitations, 50 points or 100% means complete activity limitation,Mean duration of the test: 3 to 7.8 minutes some benchmarks can be found in literature, Vernon and Moir presented the following interpretation: 0-4points (0-8%) no disability. 5-14points (10-28%) mild disability. 15-24points (30-48%) moderate disability. 25-34points (50-64%) severe disability. 35-50points (70-100%) complete disability.
Assessing the change in Pain Pressure Threshold | Baseline and 4 weeks post-intervention
  assessment via using Pressure algometer: Pain Pressure Threshold (PPT) was measured by an algometer using a 1 cm2 disk surface area pressed vertically on MTrP. To provoke pain, pressure was increased with a speed of 1kg/cm2/s-1
Assessing the change in frequency of headache | Baseline and 4 weeks post-intervention
  Headache frequency assessed after and before 12 sessions. It was defined as the number of headache days per week. The frequency of days with headache in the past weeks was registered by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Prof Abeer Yamany, Professor, Principal Investigator — Cairo University; Dr Mariam Omran, Lecturer, Study Director — Cairo University
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No